CLINICAL TRIAL: NCT06769737
Title: The Prolonged Effects of Spinal Dexmedetomidine Versus Intravenous Dexmedetomidine on Spinal Anesthesia With Isobaric Bupivacaine: A Comparative Study
Brief Title: The Prolonging Effect of Dexmedetomidine on Spinal Anesthesia Through Different Routes if Administrations
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz Medical City (Other Government)
Responsible Party: Principal Investigator, Hebah Musalem, Anesthesia Assistant consultant, King Abdulaziz Medical City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ICTR24/001/11
Record Dates: First submitted 2024-12-02; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Spinal Anesthesia Evaluation
Keywords: dexmedetomedine; intrathecal dexmedetomedine; intravenous dexmedetomedine; spinal anesthesia prolongation

STUDY DESIGN:
Intervention Model Description: This prospective, single-blinded, randomized clinical trial compares the effects of intrathecal (IT) dexmedetomidine combined with isobaric bupivacaine and intravenous (IV) dexmedetomidine combined with intrathecal isobaric bupivacaine on the duration of spinal anesthesia. The study includes one control group and two interventional groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Controlled (No Intervention): Group A: Control group. Receiving plain isobaric "Bupivacaine 0.5%", "Bucaine®," (2.4 ml) + 0.15 ml of normal saline (placebo), total volume = 2.4 ml.
  Through IV, 15 ml of normal saline ( placebo) will be received over 30 mins.
- Dexmedetomidine HCL IT (Experimental): Group B: RECEIVING IT "Dexmedetomidine HCL," "Demexa®," Through IT, receiving plain isobaric "Bupivacaine 0.5%", "Bucaine®," (2.4 ml) +3mcg of "Dexmedetomidine HCL, (0.15 ml), total volume = 2.4 ml.
  Through IV, 15 ml of normal saline ( placebo) will be received over 30 mins.
  Interventions: Drug: Interventional group#1
- Dexmedetomidine HCL IV (Experimental): Group C: RECEIVING IV "Dexmedetomidine HCL," "Demexa®,"
  Through IT, receiving plain isobaric "Bupivacaine 0.5%", "Bucaine®," (2.4 ml) + Placebo of normal saline (0.15 ml), total volume = 2.4 ml.
  Through IV, 0.5 mcg/kg of "Dexmedetomidine HCL" is prepared in a concentration of 2 mcg/ml ( maximum of 15 ml, 30 mcg) over 30 mins.
  Interventions: Drug: Interventional group#2

INTERVENTIONS:
Drug: Interventional group#1 — The intrathecal mixture of spinal anesthesia: 12 mg of isobaric "Bupivacaine 0.5%", "Bucaine®," (2.4 ml) + 20 mcg of "Fentanyl," "Martindale pharma Fentanyl®," 50mcg/ml (0.4ml) + 3 mcg of "Dexmedetomidine HCL," "Demexa®," 4mcg/ml (0.75 ml) total volume = 3.55 ml.
  The Bromage score will be assessed by the anesthesiologist every 5 minutes after positioning the patient supine until the first incision. The Bromage score is a clinical scale used to determine motor block during regional anesthesia by evaluating lower limb movement: Grade 0: Full movement of hips, knees, and ankles (no block). Grade 1: Unable to lift the leg but can move knees and ankles (partial block). Grade 2: Unable to bend the knee but can move ankles (near-complete block). Grade 3: No movement in hips, knees, or ankles (complete block). Dermatomal coverage will be assessed simultaneously till it reaches the L1-L2 level. Also, The Ramsay Sedation Scale (RSS) will be used to evaluate the sedation depth, if any.
  Other Names: Intrathecal "Dexmedetomidine HCL," "Demexa®,"
  Arms: Dexmedetomidine HCL IT
Drug: Interventional group#2 — The intrathecal mixture of spinal anesthesia: 12 mg of isobaric "Bupivacaine 0.5%", "Bucaine®," (2.4 ml) + 20 mcg of "Fentanyl," "Martindale pharma Fentanyl®," 50mcg/ml (0.4ml) total volume = 2.8 ml.
  The intravascular mixture consists of 0.5 mcg/kg of "Dexmedetomidine HCL," "Demexa®," and a maximum of 30 mcg diluted to 4 mcg/ml. According to body weight, the total volume is 7.5 ml or less and given using a syringe pump over 30 minutes. The anesthesiologist will start the infusion once the patient is positioned supine post-spinal anesthesia and has stable hemodynamics. The Bromage score will be assessed by the anesthesiologist every 5 minutes after positioning the patient supine until the first incision reaches grade 3: No movement in hips, knees, or ankles (complete block). The anesthesiologist will assess dermatomal coverage until it reaches the L1-L2 and calculate the Ramsay Sedation Scale (RSS) of the depth of sedation aiming for level 2: Patient is cooperative, oriented, and calm
  Other Names: Intravascular "Dexmedetomidine HCL," "Demexa®,"
  Arms: Dexmedetomidine HCL IV

SUMMARY:
This prospective, double-blinded, randomized clinical trial aims to examine the effects of combining isobaric bupivacaine with dexmedetomidine administered intrathecally (IT), compared to the combination of isobaric bupivacaine administered intrathecally and dexmedetomidine administered intravenously (IV), on spinal anesthesia prolongation time in minutes, time of regression from Bromage score 3 to 0.

DETAILED DESCRIPTION:
Dexmedetomidine, an α2-adrenergic agonist, is commonly used in anesthetic practice for various applications, including premedication, as an adjunct to general anesthesia, sole anesthetic agent, and sedation in intensive care settings. Its effects include enhancing the efficacy of other anesthetic drugs, inducing perioperative sympatholysis, and lowering blood pressure by stimulating central α2 and imidazoline receptors.

Spinal anesthesia is a type of regional anesthesia that involves administering a local anesthetic directly into the cerebrospinal fluid surrounding the spinal cord and nerve roots. It is primarily used for procedures below the umbilicus, such as orthopedic surgeries involving joints and bones.

The 0.5% isobaric formulation of bupivacaine is characterized by a slower onset compared to hyperbaric formulations but provides a longer duration of both sensory and motor blockade. Achieving successful spinal anesthesia (SA) depends on selecting the appropriate dose of isobaric bupivacaine. Administering an excessive dose can lead to high spinal anesthesia, while an insufficient dose may result in inadequate cephalad spread.

A retrospective observational study involving 1,079 adult patients who received spinal anesthesia with 0.5% isobaric bupivacaine between 2018 and 2021 investigated the relationship between the bupivacaine dose and block height. The study concluded that for patients younger than 60 years, doses of 15-17 mg (3.0-3.4 mL) were optimal, while doses of 10.5-16 mg (2.1-3.2 mL) were suitable for patients aged 60 years or older. These doses achieved a T5-T10

Over the years, various agents have been combined with local anesthetics (LA) to extend the duration of action in both spinal anesthesia via intrathecal (IT) administration and peripheral nerve blocks (PNB), achieving varying levels of success. Dexmedetomidine, a highly selective α2-adrenergic receptor agonist, offers several advantages as an adjuvant. These include its sedative and analgesic effects (acting at both spinal and supraspinal levels), anti-anxiety properties, inhibition of sympathetic activity, mild respiratory depression, and hemodynamic stability.

Intrathecal α2-adrenergic receptor agonists, including dexmedetomidine, have been shown to exhibit antinociceptive properties for both somatic and visceral pain. Studies using small doses of intrathecal dexmedetomidine (e.g., 3 µg) in combination with bupivacaine for spinal anesthesia demonstrated faster motor block onset, prolonged motor as well as sensory block durations, and preserved hemodynamic stability without causing significant sedation.

The dose-dependent effects of dexmedetomidine have been extensively studied. Randomized clinical trials (RCTs) comparing doses (e.g., 3 µg vs. 5 µg with isobaric Ropivacaine and 5 µg vs. 10 µg with isobaric bupivacaine) consistently concluded that higher doses of dexmedetomidine enhanced the onset and prolonged the duration of sensory and motor block when used as an adjuvant in spinal anesthesia.

Intravenous dexmedetomidine has also been shown to prolong the sensory and motor block of bupivacaine through its supraspinal anesthetic and analgesic actions. However, its intravenous administration is associated with a dose-dependent risk of bradycardia. A systematic review and meta-analysis conducted in 2013, which included 364 patients from seven randomized controlled trials of intermediate to high quality, examined the effects of intravenous dexmedetomidine on spinal anesthesia duration. The analysis found that motor block duration increased by approximately 21% (P < 0.00001). Importantly, no significant differences in the incidence of hypotension or postoperative sedation were observed between the dexmedetomidine and placebo groups, and none of the patients experienced respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients in adult age group more than 18 years old
* ASA classification I, II, and III.
* Orthopedic surgery, including total hip replacement (THR) and total knee replacement (TKR).
* No history of Obstructive sleep apnea

Exclusion Criteria:

* Patient below 18 years old of both genders.
* ASA classification of IV and more.
* Patients with a height of less than 150 cm.
* Patients on alpha-two antagonist ACE inhibitors and CCB.
* Patient received intrathecal morphine, intravascular dexamethasone, or Midazolam
* Patient who can't tolerate fluid challenge. Example: ESRD, HF…etc.
* Any contraindication for neuraxial procedure. Examples: coagulopathy, severe AS, sepsis…etc.
* Psychiatric patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Regression time of Bromage score from 3 to 0 | Patients' recruitment and participation in the study will be over 3-4 month, as the load of lower limb surgery at KAMC is high. Subjects' participation will be throughout the surgery time and 45 mins later in PACU if there was not a reason for delay.
  This double-blind study will include 75 participants divided equally into three groups: A, B, and C. The IT medication injection / IV infusion start time is considered time zero. The Bromage score will be assessed at the motor block's onset, representing a Bromage score of 3, recorded in minutes. The record of the time to reach Bromage 3 represents the spinal anesthesia's onset time.
  The Bromage scale is a clinical scale used to determine motor block during regional anesthesia. It evaluates lower limb movement, grade 0, no motor block, to grade 3, complete motor block.
  Bromage 0; the patient can move hip, knee, and ankle. No motor block Bromage 1: the patient cannot move the hip but can move the knee and ankle. Partial block Bromage 2: the patient cannot move the hip and knee but can move the ankle. partial block Bromage 3: the patient cannot move the hip, knee, and ankle. Complete motor block A Bronage score regression to 0 during a PACU stay will represent a spinal anesthesia offset

SECONDARY OUTCOMES:
Hypotension, bradycardia and desaturation with dermatome coverage <T4 or >T4, checked by Ice test. | Patients' recruitment and participation in the study will be over 3-4 month, as the load of lower limb surgery at KAMC is high. Subjects' participation will be throughout the surgery time and 45 mins later in PACU if there was not a reason for delay.
  Investigators will monitor the side effects associated with each route of administration through close hemodynamic monitoring for heart rate (HR) in Beat per minute (BPM), Oxygen saturation (SpO2) presented in percentage (%), and blood pressure (BP) presented in millimeter mercury (mmHg), aiming for HR above 50 bpm, oxygen saturation >94%, and BP 15% around the patient's baseline blood pressure. All data will be recorded on the data collection sheet.
  To differentiate high spinal-related hemodynamic instability ( dermatome >4) versus dexmedetomidine (dermatome less than T4), the sensory block level will be checked with an ICE test, where the dermatomal coverage will be checked along the midaxillary line with an ice bag, as nipple line is representing dermatome T4.
  HR limits: 60 to 100 bpm. Lower bradycardia, higher tachycardia. BP limits, systolic 100 - 120 mmHg. Lower hypotension, higher hypertension. SpO2 limit: 100-94%, 100% standard, <94% desaturation.
Sedation score using Ramsay sedation score, aiming for score 2; calm and oriented. | Patients' recruitment and participation in the study will be over 3-4 month, as the load of lower limb surgery at KAMC is high. Subjects' participation will be throughout the surgery time and 45 mins later in PACU if there was not a reason for delay.
  The Investigators will check the Ramsay Sedation Scale (RSS) throughout the procedure. It is used to evaluate the depth of sedation in patients and divided into six scales (from scale no.1, anxious to scale no.6, no response), aiming for scale no.2: cooperative, oriented, and calm. All data will be recorded on the data collection sheet every 10 minutes for the first hour of "Dexmedetomidine" administration and 45 minutes in PACU.
  The scale is getting worse while the moving up in the scale Score 1: anxious, agitated, and restless. Score 2: Cooperative-oriented and tranquil. Score 3: The patient responds to commands only. Score 4: The patient responds to a brisk response to a light glabellar tap or loud auditory stimulation.
  Score 5: Patient sluggishly responds to a light glabellar tap or loud auditory stimulus.
  Score 6: The patient exhibits no response.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Data interpretation, analysis, and results
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Abdallah FW, Abrishami A, Brull R. The facilitatory effects of intravenous dexmedetomidine on the duration of spinal anesthesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jul;117(1):271-8. doi: 10.1213/ANE.0b013e318290c566. Epub 2013 Apr 30. PMID 23632057
- [Background] Kaya FN, Yavascaoglu B, Turker G, Yildirim A, Gurbet A, Mogol EB, Ozcan B. Intravenous dexmedetomidine, but not midazolam, prolongs bupivacaine spinal anesthesia. Can J Anaesth. 2010 Jan;57(1):39-45. doi: 10.1007/s12630-009-9231-6. Epub 2009 Dec 29. PMID 20039221
- [Background] Al-Mustafa MM, Abu-Halaweh SA, Aloweidi AS, Murshidi MM, Ammari BA, Awwad ZM, Al-Edwan GM, Ramsay MA. Effect of dexmedetomidine added to spinal bupivacaine for urological procedures. Saudi Med J. 2009 Mar;30(3):365-70. PMID 19271064
- [Background] Kanazi GE, Aouad MT, Jabbour-Khoury SI, Al Jazzar MD, Alameddine MM, Al-Yaman R, Bulbul M, Baraka AS. Effect of low-dose dexmedetomidine or clonidine on the characteristics of bupivacaine spinal block. Acta Anaesthesiol Scand. 2006 Feb;50(2):222-7. doi: 10.1111/j.1399-6576.2006.00919.x. PMID 16430546
- [Background] Lundblad M, Trifa M, Kaabachi O, Ben Khalifa S, Fekih Hassen A, Engelhardt T, Eksborg S, Lonnqvist PA. Alpha-2 adrenoceptor agonists as adjuncts to peripheral nerve blocks in children: a meta-analysis. Paediatr Anaesth. 2016 Mar;26(3):232-8. doi: 10.1111/pan.12825. Epub 2015 Dec 16. PMID 26671834
- [Background] Visavakul O, Leurcharusmee P, Pipanmekaporn T, Khorana J, Patumanond J, Phinyo P. Effective Dose Range of Intrathecal Isobaric Bupivacaine to Achieve T5-T10 Sensory Block Heights for Elderly and Overweight Patients: An Observational Study. Medicina (Kaunas). 2023 Mar 1;59(3):484. doi: 10.3390/medicina59030484. PMID 36984485
- [Background] Uppal V, Retter S, Shanthanna H, Prabhakar C, McKeen DM. Hyperbaric Versus Isobaric Bupivacaine for Spinal Anesthesia: Systematic Review and Meta-analysis for Adult Patients Undergoing Noncesarean Delivery Surgery. Anesth Analg. 2017 Nov;125(5):1627-1637. doi: 10.1213/ANE.0000000000002254. PMID 28708665
- [Background] Taye MG, Molla A, Teshome D, Hunie M, Kibret S, Fentie Y, Temesgen N, Engidaw MT, Fenta E. Predictors of hypoxemia after general anesthesia in the early postoperative period in a hospital in Ethiopia: an observational study. Multidiscip Respir Med. 2021 Dec 1;16(1):782. doi: 10.4081/mrm.2021.782. eCollection 2021 Jan 15. PMID 35003732
- [Background] Bekker AY, Kaufman B, Samir H, Doyle W. The use of dexmedetomidine infusion for awake craniotomy. Anesth Analg. 2001 May;92(5):1251-3. doi: 10.1097/00000539-200105000-00031. No abstract available. PMID 11323355
- [Background] Khan ZP, Ferguson CN, Jones RM. alpha-2 and imidazoline receptor agonists. Their pharmacology and therapeutic role. Anaesthesia. 1999 Feb;54(2):146-65. doi: 10.1046/j.1365-2044.1999.00659.x. PMID 10215710